CLINICAL TRIAL: NCT05314075
Title: Determination of Core Body Temperature in Parturient Warmed With Upper or Underbody Forced Air Cover (Bair Hugger)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20024184
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cesarean Section
Keywords: Thermoregulation; Forced air warming; upper or lower body forced air cover; core body temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper Body (Active Comparator)
  Interventions: Procedure: Upper Body Forced Air Warming device
- Under body (Active Comparator)
  Interventions: Procedure: Under Body Forced Air Warming device

INTERVENTIONS:
Procedure: Upper Body Forced Air Warming device — Patients will have the Bair Hugger placed over the body
  Other Names: Bair Hugger
  Arms: Upper Body
Procedure: Under Body Forced Air Warming device — Patients will have the Bair Hugger placed under the body
  Other Names: Bair Hugger
  Arms: Under body

SUMMARY:
This study is intended to calculate the core body temperature in patients who are having a Cesarean Section (C/S) and are kept warm with an Upper Body Forced Air Warming device (Bair Hugger) or underbody forced air warmer. These warming devices are approved and are a required item in many if not all surgical procedures. They are used daily throughout the hospital. The research question is: Where is the best place to position the warming blanket in pregnant mothers undergoing Cesarean section delivery. The researchers hope to compare post - operative core body temperatures in patients getting an Upper Body forced air device versus those getting an Underbody Body forced air warming device.

ELIGIBILITY:
Inclusion Criteria:

* Age =/> 18 years
* Elective non-emergent C-section

Exclusion Criteria:

* BMI<18/>40
* Bleeding Disorders e.g. hemophilia, coagulation abnormality, clotting disorders, bleeding diathesis
* Perioperative hemorrhage >1500ml
* Non-Singleton Pregnancies
* Complicated Pregnancy (e.g. Eclampsia, Pre-eclampsia)
* Conversion to Emergency C-section
* Endocrine Pathology- e.g. Thyroid Disease, Insulin Dependent Diabetes
* Inmates

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant females
Enrollment: 124 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Core body temperature | 1 hour post surgery
  Maternal core temperatures will be measured using a temperature sensing Foley catheter

CONTACTS AND LOCATIONS:
Overall Officials: Fatoumata Kromah, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No